CLINICAL TRIAL: NCT03087682
Title: Pituitary Gland Enlargement Was First Diagnosed by OCT Before There Were Any Changes at All in the Computerized and Automated Eighty Degrees Peripheral Visual Fields
Brief Title: Pituitary Gland Enlargement Was First Diagnosed by Optical Coherence Tomography (OCT)
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Dr. S.S. Michel Clinic (Other)
Responsible Party: Principal Investigator, Dr. Shawkat Michel, Principal Investigator, Dr. S.S. Michel Clinic
Other Study IDs: Pituitary gland enlargement
Record Dates: First submitted 2017-03-12; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Pituitary Mass; Diagnoses Disease
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) — OCT is used to measure thickness (numbers) of retinal nerve fibres in different areas of the retina

SUMMARY:
OCT is now an established way to measure the thickness of the Retinal Nerve Fiber Layer (RNFL) in the retina of the eye. The thickness of the RNFL is always a reflection of the number of the RNFs in any particular area of the retina. Each single RNF runs a long course starting from the cell body which is the retinal ganglion cell in the retina and ends in the thalamus of the brain where it relays visual information to other nerve cell in the thalamus. Along this long course RNFs are in close anatomical relationship with the pituitary gland crossing just above this gland about midway along their course. Hence enlargement of this gland can interfere with the RNFs.

DETAILED DESCRIPTION:
The inferior chiasmal syndrome is known to be caused by pituitary gland enlightenment because the pituitary gland lies just below the optic chiasma. The visual RNFs are organized in a very specific way along their long course from the retina to the Lateral Geniculate Body (LGB) in the thalamus. Pituitary enlargement would compromise particular RNFs. It is well known and established that pituitary enlargement, if not properly treated in time, would possibly cause bitemporal hemianopia due to interference with the crossing RNFs of the nasal half of each retina. In this study pituitary enlargement was suspected by OCT findings while the patient still had perfect peripheral visual field in each eye.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients with frequent or persistent headache of unknown reasons.

Exclusion Criteria:

* patients who were previously diagnosed with or treated from pituitary enlargement

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient who presents with frequent or persistent headache of unknown reason.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-03-15 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Thinning of the retinal nerve fibers (RNF) that are nearest to the pituitary gland, measured in micro-millimeters in OCT, were the first indication of possible enlargement of this gland. | through study completion, an average of one year.
  Pituitary gland enlargement if not treated in time can have devastating effects on vision. Early diagnosis and treatment of this problem can not be over stressed. This study describes thinning of particular RNF in each eye that led to the suspicion of pituitary enlargement and was an early sign of the inferior chiasmal syndrome. Imaging studies were used to validate the suspected result.

CONTACTS AND LOCATIONS:
Overall Officials: Shawkat S Michel, FRCS Ed, Principal Investigator — Dr. S.S. Michel Clinic
Locations (1):
- Dr. S.S. Michel Clinic, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No